CLINICAL TRIAL: NCT01100567
Title: EFFECT OF BIOMECHANICAL STIMULATION ON SKELETAL HEALTH IN ADOLESCENT AND YOUNG WOMEN WITH ANOREXIA NERVOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amy DiVasta, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-10-0461
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Anorexia Nervosa
Keywords: skeletal health; bone turnover; bone geometry; malnutrition
MeSH Terms: conditions — Anorexia Nervosa; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo platform (Placebo Comparator): Randomized to stand on placebo platform for 10 minutes/day
  Interventions: Device: Low-magnitude mechanical stimulation platform
- Low-magnitude mechanical stimulation (Active Comparator): Randomized to stand on LMMS platform 10 minutes/daily
  Interventions: Device: Low-magnitude mechanical stimulation platform

INTERVENTIONS:
Device: Low-magnitude mechanical stimulation platform — Low-magnitude mechanical stimulation platform

SUMMARY:
This study will evaluate the effects of a novel, non-pharmacologic intervention for the prevention of deleterious changes in bone density and strength in adolescents with anorexia nervosa (AN), a disease commonly treated with extended periods of bed rest and immobilization. The primary focus of the trial is to conduct a prospective short-term intervention to prevent an uncoupling of bone turnover in inpatients hospitalized for AN, and to determine the long-term effects of a biomechanical intervention on skeletal health in ambulatory adolescents with AN.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-25 years
* Diagnosis of anorexia nervosa based on DSM-IV criteria
* Female gender
* English-speaking

Exclusion Criteria:

* • Concomitant chronic diseases which affect bone health, such as cystic fibrosis, inflammatory bowel disease, celiac disease, renal disease, or diabetes mellitus

  * Use of medications known to affect bone metabolism in the last 3 months, such as:

    * Glucocorticoid therapy (including inhaled steroids)
    * Anticonvulsants
    * Combined estrogen/progestin contraceptive agents (oral contraceptive pills)
  * Depot medroxyprogesterone (Depo-Provera) use in the last 12 months
  * Current pregnancy

Ages: 11 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2009-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D DiVasta, MD, MMSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] DiVasta AD, Stamoulis C, Rubin CT, Gallagher JS, Kiel DP, Snyder BD, Gordon CM. Low-Magnitude Mechanical Signals to Preserve Skeletal Health in Female Adolescents With Anorexia Nervosa: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2441779. doi: 10.1001/jamanetworkopen.2024.41779. PMID 39480424
- [Derived] Lin JA, Stamoulis C, DiVasta AD. Associations between nutritional intake, stress and hunger biomarkers, and anxiety and depression during the treatment of anorexia nervosa in adolescents and young adults. Eat Behav. 2023 Dec;51:101822. doi: 10.1016/j.eatbeh.2023.101822. Epub 2023 Oct 26. PMID 38504970

RESULTS

PARTICIPANT FLOW:
Groups:
- LMMS: Randomized to 10 min LMMS daily
- Placebo: Randomized to sham platform 10 min daily
Period: Overall Study
Arm/Group | LMMS | Placebo
Started | 50 | 51
Completed | 38 | 35
Not Completed | 12 | 16
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Early Hospital Discharge | 6 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Deemed ineligible after consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMMS | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (2.1) | 16.2 (1.8) | 16.3 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41
BMI Z-score [Mean (Standard Deviation); unit: Z-score] | -2.34 (1.6) | -3.24 (2.66) | -2.79 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in C-telopeptides
Time Frame: Baseline to 5 days
Measure: Mean (95% Confidence Interval); unit: ng/mL/day
Arm/Group | LMMS | Placebo
Number analyzed (Participants) | 20 | 21
ng/mL/day | 0.083 [0.006 to 0.159] | -0.027 [-0.119 to 0.065]

2. Secondary Outcome: Change From Baseline in Bone Specific Alkaline Phosphatase
Time Frame: baseline to 5 days
Measure: Mean (95% Confidence Interval); unit: ug/L/day
Arm/Group | LMMS | Placebo
Number analyzed (Participants) | 20 | 21
ug/L/day | -0.07 [-0.26 to 0.14] | -0.36 [-0.68 to -0.04]

ADVERSE EVENTS:
Arm/Group | LMMS | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No